CLINICAL TRIAL: NCT03599180
Title: Clinical Research Protocol of Systematic Biology Mechanism for Sensitized Acupoint Micro-physicochemical Environment Changes in Knee Osteoarthritis Patients
Brief Title: Clinical Protocol of Sensitized Acupoint Changes in Knee Osteoarthritis Patients
Status: Completed | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: 81590953
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2018-06

CONDITIONS: Microdialysis
Keywords: Knee Osteoarthritis; Sensitized Acupoints; Microdialysis; High performance liquid chromatography（HPLC）
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Microdialysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — microdialysate of KOA patients' sensitised acupoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Knee Osteoarthritis group: KOA patients without accept treat in the past month
  Interventions: Device: microdialysis
- Control group: Heathly volunteers
  Interventions: Device: microdialysis

INTERVENTIONS:
Device: microdialysis — Use microdialysis skill to collect dialyzate at sensitization acupoints

SUMMARY:
Based on the research background and the preliminary research basis of the research group, in order to answer the material basis and micro-physical environment change characteristics of knee osteoarthritis sensitization acupoints and provide scientific basis for in-depth study of sensitization of acupoints. This study plans to use knee osteoarthritis as a research vehicle, and use microdialysis combined with high performance liquid chromatography to analyze the local material basis and key indicators of common sensitization points in knee osteoarthritis.

DETAILED DESCRIPTION:
This trial is a single-centre, normal controlled, parallel group, clinical trial. The trial is an explorative, pilot trial designed to reveal the change of the main material group in sensitized acupoints caused by knee osteoarthritis, and provide the key signal substance and its changing characteristics of knee osteoarthritis sensitized acupoints.

ELIGIBILITY:
Inclusion Criteria:

Meets the diagnosis criteria of knee osteoarthritis. Age between 45 and 70 years. Meets imaging examination X-ray Kellgren and Laerence classification standards grade I-III.

Patients who meet the criteria for early or mid-term stage of knee osteoarthritis.

Discontinue use of pain medications and hormone drugs during the trial. The patient's vital signs are stable, can read his own medical history, and can cooperate with the relevant examination and treatment.

Signed the informed consent voluntarily.

Exclusion Criteria:

Seriously patients with surgical indications Associated systemic arthropathies, e.g. rheumatoid arthritis and gout Heart failure Bleeding diathesis Liver failure knee arthroplasty There are diseases that may seriously endanger life, such as cardiovascular and cerebrovascular diseases, renal and liver failure, hematopoietic system diseases, etc.

Patients with mental illnesses that cannot be completed or are not suitable for treatment and examination Patients who received treatment including traditional Chinese medicine, western medicine, acupuncture, massage and physiotherapy within the past month Patients on steroids History of intra articular injection of steroid within last six months Joint irrigation or arthroscopy has been performed within the past year Have had knee arthroplasty At the same time participate in other studies

Ages: 38 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 32 KOA patients and 32 normal volunteers will be included
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Serotonin concentration | 2018-7-12---2020-7-1
  The serotonin concentration of KOA patients' sensitized acupoints was compared with that of the normal acupoints in healthy volunteers.

SECONDARY OUTCOMES:
Histamine concentration | 2018-7-12---2020-7-1
  The histamine concentration of KOA patients' sensitized acupoints was compared with that of the normal acupoints in healthy volunteers.
Adenosine triphosphate concentration | 2018-7-12---2020-7-1
  The adenosine triphosphate concentration of KOA patients' sensitized acupoints was compared with that of the normal acupoints in healthy volunteers.
WOMAC score | 2018-7-12---2020-7-1
  The WOMAC score of KOA patients was compared with healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shuguang, Bachelor, Study Director — No.39,Shi'er Qiao road,Jinniu district, Chengdu, Sichuan province, China
Locations (1):
- Shuguang, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li S, Chai XN, Zuo CY, Lv P, Tang Y, Tan HJ, Liu LZ, Yin HY, Yu SG. Metabolic profiling of dialysate at sensitized acupoints in knee osteoarthritis patients: A study protocol. Medicine (Baltimore). 2019 Nov;98(45):e17843. doi: 10.1097/MD.0000000000017843. PMID 31702640